CLINICAL TRIAL: NCT04621500
Title: Vitamin D Supplementation in RNA-seq Profiles of Single-core Prostate Samples, Including Diversity and Stress Determinants, Among Veterans
Brief Title: Vitamin D Supplementation in RNA-seq Profiles of Single-core Prostate Samples, Among Veterans
Acronym: VitD/RNA-seq
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Ralph H. Johnson VA Medical Center (U.S. Federal Agency); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00085140; 5U54MD010706-03 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-11-09 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Vitamin D Deficiency; Stress Reaction
MeSH Terms: conditions — Prostatic Neoplasms; Vitamin D Deficiency; Fractures, Stress | interventions — Cholecalciferol; RNA-Seq; Allostasis

STUDY DESIGN:
Intervention Model Description: Single, open-label group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label (Other): All enrolled subjects will receive vitamin D3 at 4,000 IU daily for approximately one year.
  Interventions: Drug: cholecalciferol; Procedure: Standard of Care Prostate Biopsy - collection of 13th core for RNA-seq; Procedure: Standard of Care Prostate Biopsies at baseline and after one year vitamin D3 supplementation; Diagnostic Test: Allostatic Load

INTERVENTIONS:
Drug: cholecalciferol — Enrolled subjects will supplement with vitamin D3 at 4,000 IU daily for one year
  Other Names: vitamin D3
Procedure: Standard of Care Prostate Biopsy - collection of 13th core for RNA-seq — RNA-seq analysis will be used to (a) identify changes in transcriptional profiles and biological pathways in the prostate between African American and Caucasian men and (b) compare Allostatic Load results to determine stress response and (c) identify changes in the molecular signature in relation to vitamin D levels
Procedure: Standard of Care Prostate Biopsies at baseline and after one year vitamin D3 supplementation — Pathology results of the prostate biopsies will be analyzed for changes in the (a) Gleason Score (b) the number of positive cores (0 to 12) and (c) the highest percentage of positive core involvement (0 to 100%).
Diagnostic Test: Allostatic Load — Diagnostic Test: Allostatic Load Measurements at baseline and after one year vitamin D3 supplementation Allostatic Load measurements to determine body stress compared at baseline and after one year of vitamin D3 supplementation. Also compared with RNA-seq results to determine stress response.
  Other Names:
  Bloodwork for HgbA1c, lipid profile, creatinine, albumin and vitamin D levels. Body measurements: Ht. Wt, BMI, waist and hip measurements for waist/hip ratio. Measurements of systolic and diastolic blood pressure and heart rate

SUMMARY:
Veterans between the ages of 50-75, who are having a prostate biopsy, will be recruited for their permission to collect an extra biopsy core for RNA-sequencing. If the participants' treatment decision is Active Surveillance, they will be enrolled into the intervention phase of the study. They will receive supplementation with Vitamin D3 (4,000 IU) daily with repeat (surveillance) prostate biopsy one year later. At that time an extra prostate sample core will be collected for RNA-sequencing to determine changes over time. Measurements for allostatic load (body stress/inflammatory markers) will also be collected at the time of enrollment and at the repeat prostate biopsy visit.

DETAILED DESCRIPTION:
This is an open-label pilot study. The goal is to investigate the transcription and biological pathways in prostate cancer that are especially relevant to prostate cancer disparities between African American and Caucasian men. Also, to determine any significant differences in the molecular signature that exist in African American and Caucasian men in relation to their Vitamin D levels.

Recruitment will be at the Urology Clinic at the Ralph H. Johnson VA Medical Center in Charleston, SC. Men who are scheduled for a Standard of Care prostate biopsy will be consented for their permission to collect an extra prostate tissue core for RNA-sequencing.

After the pathology report is discussed by their Urologist, and the treatment decision is Active Surveillance, the participant is enrolled into the Intervention Phase. At that time, baseline allostatic load measurements (Blood pressure, pulse, waist/hip ratio, height, and weight for BMI) and bloodwork: (lipid panel, HgbA1c, albumin and creatinine, IL-6, CRP, and DHEA-s (inflammatory markers) plus a Vitamin D level, will be collected. Vitamin D3 soft gels (4,000 IU) daily (six months' supply) will be dispensed. A Social Determinants survey will also be dispensed for subject completion.

At the Urology Standard of Care six-month follow-up appointment, the vitamin D serum level will be collected and the next six months' supply of vitamin D3 will be dispensed.

At the Urology Standard of Care follow-up (repeat at 1 year) surveillance prostate biopsy, an extra prostate tissue core will be collected for RNA-sequencing. The allostatic load measurements and bloodwork will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

Recruitment:

* scheduled for prostate biopsy
* permission for investigators to follow subject's post biopsy diagnosis, treatment decision and follow-up care (including subsequent prostate biopsies).

Enrollment:

* diagnosis of prostate cancer
* treatment recommendation or subject decision of Active Surveillance
* agreement to supplement with vitamin D3 4,000 IU daily for approximately one year
* standard of care repeat PSA at six months and surveillance prostate biopsy at one year

Exclusion Criteria:

* current vitamin D3 supplementation > 2,000 IU daily
* inability or unwillingness to continue to participate in the study

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals having a prostate biopsy are eligible for recruitment.
Enrollment: 60 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chanita Hughes-Halbert, PhD, Study Director — MUSC Psychiatry and Behavioral Sciences
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in the urology clinic at the Ralph H. Johnson VAMC. All patients who were eligible for active surveillance for prostate cancer were offered enrollment and were followed at the same location. They were recruited from 6/4/19 until 2/4/22
Groups:
- Open Label: All enrolled subjects will receive vitamin D3 at 4,000 IU daily for approximately one year.
  cholecalciferol: Enrolled subjects will supplement with vitamin D3 at 4,000 IU daily for one year
  Standard of Care Prostate Biopsy - collection of 13th core for RNA-seq: RNA-seq analysis will be used to (a) identify changes in transcriptional profiles and biological pathways in the prostate between African American and Caucasian men
  Standard of Care Prostate Biopsies at baseline and after one year vitamin D3 supplementation: Pathology results of the prostate biopsies will be analyzed for changes in the (a) Gleason Score (b) the number of positive cores (0 to 12) and (c) the highest percentage of positive core involvement (0 to 100%).
Period: Overall Study
Arm/Group | Open Label
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 31
Sex: Female, Male [Count of Participants; unit: Participants] — All males
  Participants
    Female | 0
    Male | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 33
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60
Age (years) [Median (Inter-Quartile Range); unit: years] | 65 [46 to 76]
Body Mass Index (BMI) [Median (Full Range); unit: Measured in kilograms per meters squared] — Measured in kilograms per meters squared
  Measured in kilograms per meters squared | 29.2 [17.8 to 52.1]
Vitamin D (ng/ml) [Median (Full Range); unit: nanograms per milliliter] — Measured in nanograms per milliliter
  nanograms per milliliter | 28 [4.8 to 68.6]
Total cholesterol (mg/dl) [Median (Full Range); unit: milligrams per deciliter] — Measured in milligrams per deciliter
  milligrams per deciliter | 189 [85 to 271]
HbA1c level% [Median (Full Range); unit: Percentage] | 5.6 [4.1 to 10.5]
psa (mcg/l) [Median (Full Range); unit: micrograms per liter] — Measured in micrograms per liter
  micrograms per liter | 6.21 [0.56 to 31.5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Change in Transcriptional Profiles After Vitamin D Supplementation.
Description: RNA-sequencing analysis will be utilized to identify changes in transcriptional profiles and biological pathways in the prostate between African American and Caucasian men.
Time Frame: Scheduled prostate biopsy at baseline and repeat biopsy after 1 year
Population: We analyzed all subjects and compared initial biopsy results and RNA sequencing information at baseline and after supplemental vitamin D3 one year later. We looked at modifications of signaling pathways from baseline and after treatment and also compared African-Americans vs. Caucasions
Measure: Number; unit: percentage of subjects
Arm/Group | Open Label
Number analyzed (Participants) | 60
percentage of subjects | 100
Statistical Analysis 1: Comparison: Open Label; Test type: Other — The sequencing transcriptional profile cannot be analyzed by a statistical method; In this open label study, the RNA sequencing transcription analysis was performed to assess if the transcriptome would be modified by vitamin D supplementation and it uniformaly was

2. Secondary Outcome: Median Percentage of Positive Cores at 1-year Post-baseline
Description: During a routine prostate biopsy, 12 core samples are collected: 2 samples from the top right, front and back, 2 from the top left, front and back; 2 from the middle right and 2 from the middle left; 2 from the bottom right and 2 from the bottom left. When the 12 cores are examined under the microscope, the Pathologist identifies which cores contain cancer cells (or are positive for cancer).
  Therefore, the pathology report will identify the number of positive cores between 0 to 12.
  Changes to the baseline and repeat prostate biopsy positive core will be analyzed.
Time Frame: Scheduled prostate biopsy at baseline and repeat biopsy after 1 year
Measure: Median (Full Range); unit: percentage of positive cores
Arm/Group | Open Label
Number analyzed (Participants) | 60
percentage of positive cores | 0.5 [0 to 5]

3. Secondary Outcome: Identify Changes in Molecular Signature That Exist in AA and Caucasian Men in Relation to Vitamin D Levels
Description: RNA-seq analyses of prostate tissue plus allostatic load measurements to determine stress response
Time Frame: Scheduled prostate biopsies at baseline and after one year vit D supplementation plus allostatic load measurements at baseline and one yeat visits
Population: Number of positive cores per patient on a standard prostate biopsy involving systematic sampling of the prostate.
Measure: Mean (99% Confidence Interval); unit: number of positive cores
Arm/Group | Open Label
Number analyzed (Participants) | 60
number of positive cores | 17.4 [16.336 to 18.464]

ADVERSE EVENTS:
Time Frame: throughout the study, up to 2 years and 8 months
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT04621500/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT04621500/ICF_000.pdf